CLINICAL TRIAL: NCT00048165
Title: A Double-Blind, Placebo -Controlled, Randomized Study to Assess the Efficacy and Safety of Zenapax in Combination With CellCept, Cyclosporine, and Corticosteroids in Patients Undergoing Cardiac Transplantation.
Brief Title: A Study to Evaluate the Efficacy and Safety of Zenapax in Combination With CellCept, Cyclosporine, and Corticosteroids in Patients Undergoing Cardiac Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NR15880
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Daclizumab; Methylprednisolone; Mycophenolic Acid; Cyclosporine

ARMS (2):
- Daclizumab (Experimental): Daclizumab will be administered as a intravenous dose of 1 milligrams per kilogram [mg/kg] on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID], cyclosporine 1-4 mg/kg IV or 2-6 mg/kg, and 500-1000 mg IV methylprednisolone peri operative switch to oral at 0.5-1 mg/kg/day followed by tapering.
  Interventions: Drug: Daclizumab; Drug: Methylprednisolone; Drug: Mycophenolate mofetil; Drug: cyclosporine
- Placebo (Placebo Comparator): Matching placebo will be administered on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID], cyclosporine 1-4 mg/kg IV or 2-6 mg/kg orally, and 500-1000 mg IV methylprednisolone peri-op switch to oral at 0.5-1 mg/kg/day followed by tapering.
  Interventions: Drug: Methylprednisolone; Drug: Mycophenolate mofetil; Drug: Placebo; Drug: cyclosporine

INTERVENTIONS:
Drug: Daclizumab — Daclizumab will be administered as 1 mg/kg IV within 12 hours post-op (Day 1), and Days 8, 22, 36 and 50.
  Other Names: Zenapax
  Arms: Daclizumab
Drug: Methylprednisolone — Methylprednisolone will be administered as 500-1000 mg IV and peri-operative switch to oral at 0.5-1 mg/kg/day followed by tapering till 0.0-0.15 mg/kg/day (up to 365 days).
Drug: Mycophenolate mofetil — Mycophenolate mofetil will be administered as 1.5 grams bid begun post-op, either IV or orally as required up to 365 days.
Drug: Placebo — Matching placebo will be administered on Days 1, 8, 22, 36, and 50.
  Arms: Placebo
Drug: cyclosporine — Cyclosporine will be administered as 1-4 mg/kg IV or 2-6 mg/kg orally up to 365 days.

SUMMARY:
The purpose of the study is to compare the number of randomized participants in each treatment group who experience an acute rejection episode in the first 6 months after undergoing cardiac transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be undergoing their first cardiac allograft transplant
* Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to transplantation
* Women of childbearing potential must use two reliable forms of contraception simultaneously. Effective contraception must be used before beginning study drug therapy, and for 4 months following discontinuation of study drug therapy
* Participants and/or their guardians must be willing and be capable of understanding risks and comply with the purpose of the study

Exclusion Criteria:

* Previous organ transplants
* Participants receiving multiple organs
* Participants requiring ventricular assist device (VAD) upon completion of transplantation surgery
* Women lactating, pregnant or of childbearing potential not using, or who are unwilling to use two reliable forms of contraception simultaneously during the study
* History of a psychological illness or condition which would interfere with the participant's ability to understand the requirements of the study
* White blood count =<2500/mm^3, platelets =<50,000/mm^3 or hemoglobin =<6 g/dL
* HIV-1, the presence of positive HBsAg, or chronic active hepatitis C
* Active peptic ulcer disease
* Severe diarrhea or other gastrointestinal disorders which might interfere with their ability to absorb oral medication
* Malignancies within the past 5 years, excluding skin carcinoma that have been adequately treated
* Participants who have received within the past 30 days or require concomitant treatment with other investigational drugs or immunosuppressive medications that are prohibited for this study
* Inability to start microemulsion form of cyclosporine within 72 hours

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (22):
  - Birmingham, Alabama
  - Los Angeles, California
  - Tampa, Florida
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Albuquerque, New Mexico
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (2):
  - London, Ontario
  - Ottawa, Ontario
- Germany (2):
  - Frankfurt am Main
  - Hanover
- Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 31 centers in four countries from 28 Aug 1999 to 19 Aug 2002.
Groups:
- Daclizumab: Eligible participants were administered an intravenous (IV) dose of daclizumab (1 milligrams per kilogram [mg/kg]) on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID]), cyclosporine (1-4 mg/kg IV or 2-6 mg/kg orally/nasogastric), and corticosteroid (methylprednisolone, 500-1000 mg IV peri-operative switch to oral at 0.5-1 mg/kg/day followed by tapering). Participants received mycophenolate mofetil, cyclosporine, and corticosteroid up to 365 days.
- Placebo: Eligible participants were administered an IV dose of matching placebo (1 milligrams per kilogram [mg/kg]) on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID]), cyclosporine (1-4 mg/kg IV or 2-6 mg/kg orally/nasogastric), and corticosteroid (methylprednisolone, 500-1000 mg IV peri-operative switch to oral at 0.5-1 mg/kg/day followed by tapering). Participants received mycophenolate mofetil, cyclosporine, and corticosteroid up to 365 days.
Period: Completed 6 Months Study
Arm/Group | Daclizumab | Placebo
Started | 216 | 218
Completed | 165 | 170
Not Completed | 51 | 48
Not completed — Administration/Other | 8 | 8
Not completed — Abnormality of laboratory test | 1 | 0
Not completed — Adverse event/intermittent illness | 14 | 11
Not completed — Death | 12 | 6
Not completed — Insufficient therapy | 1 | 4
Not completed — Other violation | 4 | 6
Not completed — Refused treatment | 5 | 5
Not completed — Violation criteria | 0 | 2
Not completed — Did not receive study drug | 6 | 6
Period: Completed 12 Months Study
Arm/Group | Daclizumab | Placebo
Started | 165 | 170
Completed | 162 | 167
Not Completed | 3 | 3
Not completed — Administration/Other | 0 | 2
Not completed — Death | 2 | 1
Not completed — Did not co-operate/Withdrew | 1 | 0

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants who were randomized into the study, whether they received the study drug or not.
Groups:
- Daclizumab: Eligible participants were administered an intravenous daclizumab (1 milligrams per kilogram [mg/kg]) on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID], cyclosporine (1-4 mg/kg IV or 2-6 mg/kg orally/nasogastric), and corticosteroid (methylprednisolone, 500-1000 mg IV pre-operative switch to oral at 0.5-1 mg/kg/day followed by tapering). Participants received mycophenolate mofetil, cyclosporine, and corticosteroid up to 365 days.
- Placebo: Eligible participants were administered an intravenous matching placebo on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID], cyclosporine (1-4 mg/kg IV or 2-6 mg/kg orally/nasogastric), and corticosteroid (methylprednisolone, 500-1000 mg IV pre-operative switch to oral at 0.5-1 mg/kg/day followed by tapering). Participants received mycophenolate mofetil, cyclosporine, and corticosteroid up to 365 days.
- Total: Total of all reporting groups
Arm/Group | Daclizumab | Placebo | Total
Number analyzed (Participants) | 216 | 218 | 434
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.75) | 53.1 (11.89) | 52.8 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 86
  Male | 171 | 177 | 348

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Acute Rejection Episode Within 6 Months Post-Transplant
Description: The acute rejection episode was a composite end-point of acute rejection and treatment failure within 6 months post-transplant (PT). Participants with acute rejection included participants with a biopsy histology of International Society of Heart and Lung Transplant (ISHLT) Grade IIIA, IIIB, or IV and participants with hemodynamic compromise (HDC) who were treated for acute rejection (whether or not a biopsy was done and regardless of the grade of the biopsy). Participants who had treatment failure included participants who died within 6 months of transplantation before experiencing acute rejection or who were re-transplanted within 6 months of the primary transplantation and who did not experience an acute rejection or who were lost to follow-up.
Time Frame: Up to 6 months PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants | 77 | 104
Statistical Analysis 1: Comparison: Daclizumab vs Placebo; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; percent mean difference = -12.0, 95% CI 2-sided [-20.9 to -3.3]

2. Secondary Outcome: Number of Participants Who Developed Acute Rejection Episode Within the 12 Months PT
Description: The acute rejection episode was a composite end-point of acute rejection and treatment failure within 6 months. Participants with acute rejection included participants with a biopsy histology of ISHLT Grade IIIA, IIIB, or IV and participants with hemodynamic compromise (HDC) who were treated for acute rejection (whether or not a biopsy was done and regardless of the grade of the biopsy). Participants who had treatment failure included participants who died within 6 months of transplantation before experiencing acute rejection or who were re-transplanted within 6 months of the primary transplantation and who did not experience an acute rejection or who were lost to follow-up
Time Frame: Up to 12 months PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants | 97 | 116
Statistical Analysis 1: Comparison: Daclizumab vs Placebo; Test type: Superiority or Other; p = 0.063, Cochran-Mantel-Haenszel; percent mean difference = -8.6, 95% CI 2-sided [-17.7 to 0.5]

3. Secondary Outcome: Number of Acute Rejection Episodes Per Participant Within the First 6 Months and 12 Months PT
Description: The number of participants with 0,1, 2, 3 or 4 episodes at 6 and 12 months PT were reported. An episode of acute rejection was defined according to the date of positive biopsy of Grade IIIA or worse or the date of start of treatment for HDC, whichever came first.
Time Frame: Within 6 months and 12 months PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants
  Within 6 months, 0 episode | 139 | 114
  Within 6 months, 1 episode | 63 | 82
  Within 6 months, 2 episodes | 12 | 19
  Within 6 months, 3 episodes | 2 | 2
  Within 6 months, 4 episodes | 0 | 1
  Within 12 months, 0 episode | 119 | 102
  Within 12 months, 1 episode | 68 | 90
  Within 12 months, 2 episodes | 23 | 19
  Within 12 months, 3 episodes | 3 | 5
  Within 12 months, 4 episodes | 3 | 2

4. Secondary Outcome: Number of Participant Who Died Within 6 Months 12 Months and 3 Years PT
Description: The survival of the graft and participants at 6,12 months and 3 years PT was reported
Time Frame: At 6 months, 12 months , 3 years PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants
  Within 6 months | 16 | 10
  Within 12 months | 21 | 12
  Within 3 years | NA — Data was not collected | NA — Data was not collected

5. Secondary Outcome: Number of Participants With Worst ISHLT Biopsy Grade Within First 6 Months and 12 Months PT
Description: The number of participants with Worst International Society of Heart and Lung Transplant (ISHLT) grade within first 6 months and 12 months PT were reported. ISHLT is a standardized grading method to determine the acute cellular rejection on endomyocardial biopsy ; where 0= no rejection, IA= focal (perivascular or interstitial) infiltrate without necrosis, IB= diffuse but sparse infiltrate without necrosis, II=one focus only with aggressive infiltration and/or focal myocyte damage, IIIA=multifocal aggressive infiltrates and/or myocyte damage, IIIB= diffuse inflammatory process with necrosis, IV= diffuse aggressive polymorphous and/or infiltrate and/or edema and/or hemorrhage and/or vasculitis, with necrosis
Time Frame: Within 6 months and 12 months PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants
  Within 6 months, Grade 0 | 9 | 5
  Within 6 months, Grade IA | 64 | 51
  Within 6 months, Grade IB | 26 | 28
  Within 6 months, Grade II | 55 | 38
  Within 6 months, Grade IIIA | 48 | 74
  Within 6 months, Grade IIIB | 8 | 15
  Within 6 months, Grade IV | 1 | 1
  Within 12 months, Grade 0 | 7 | 4
  Within 12 months, Grade IA | 56 | 39
  Within 12 months, Grade IB | 22 | 21
  Within 12 months, Grade II | 51 | 47
  Within 12 months, Grade IIIA | 63 | 85
  Within 12 months, Grade IIIB | 11 | 15
  Within 12 months, Grade IV | 1 | 1
Statistical Analysis 1: Comparison: Daclizumab vs Placebo; Comparison of Daclizumab and Placebo for 6 months were presented; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Daclizumab vs Placebo; Comparison of Daclizumab and Placebo for 12 months were presented; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel

6. Secondary Outcome: Median Time to First Acute Rejection Episode Within the First 6 Months and 12 Months PT
Description: The median time to first acute rejection episode within first 6 months and 12 months PT was reported.
Time Frame: Within 6 months and 12 months PT
Population: The randomized population included all participants who were randomized into the study, whether they received the study drug or not. The number of participants analyzed for the specified timepoints are denoted by 'n'.
Measure: Median (Full Range); unit: days
Groups:
- Placebo: Eligible participants were administered an IV dose of matching placebo on Days 1, 8, 22, 36, and 50, along with mycophenolate mofetil (one dose of 1.5 mg twice daily [BID], cyclosporine (1-4 mg/kg IV or 2-6 mg/kg orally/nasogastric), and corticosteroid (methylprednisolone, 500-1000 mg IV pre-operative switch to oral at 0.5-1 mg/kg/day followed by tapering). Participants received mycophenolate mofetil, cyclosporine, and corticosteroid up to 365 days.
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 97 | 116
days
  Within 6 months (n= 77, 104) | 61 [2 to 210] | 21 [1 to 240]
  Within 12 months (n=97, 116) | 96 [2 to 372] | 26 [1 to 377]

7. Secondary Outcome: Number of Participants Using Monomurab Cluster of Differentiation 3, Orthoclone Polyclonal Antithymocyte Globulin or Antilymphocyte Globulin in the First 6 Months and 12 Months PT
Description: The number of participants who received monomurab Cluster of differentiation 3, orthoclone, polyclonal antithymocyte globulin or antilymphocyte globulin for treatment of biopsy proven rejection or HDC within 6 and 12 months PT were reported.
Time Frame: Within 6 months and 12 months PT
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 218
participants
  Within 6 months | 17 | 19
  Within 12 months | 23 | 21

8. Secondary Outcome: Mean Maintenance Doses of Mycophenolate Mofetil, Cyclosporine, and Cumulative Dose of Corticosteroids at 6 and 12 Months PT
Description: The maintenance doses of mycophenolate mofetil (1.5g twice a day daily), cyclosporine (1-4 mg/kg IV or 2-6 mg/kg oral [PO]/nasogastric [NG] within 72 hours post-operative]), and cumulative dose of corticosteroids (500-1000 mg IV methylprednisolone pre-operative switched to oral at 0.5-1 mg/kg/day. Tapered to 0.2 mg/kg/d by Day 28, 0.1-0.15 mg/kg/day from Days 36 to 90, and 0.1-0.15 mg/kg/day from Days 120 to 180)at 6 and 12 months PT were reported. Maintenance dose was calculated as total dose per day summed over all days that a participant was administered drug within the specified time interval, divided by number of days that a participant took drug within that time interval.
Time Frame: Within 6 months and 12 months PT
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 203 | 206
mg
  MMF dose, 6 months PT (n=193, 201) | 2522.2 (791) | 2450 (748.9)
  MMF dose,12 months PT (n=188, 194) | 2394.1 (808) | 2380.1 (779.2)
  IV Cyclosporine dose, 6 months PT (n=2, 1) | 86.11 (102.7) | 38.1 (NA) — Data not collected
  IV Cyclosporine dose, 12 months PT (n=4, 2) | 93.5 (84.3) | 46.7 (18)
  PO/NG Cyclosporine dose, 6 months PT (n=184, 182) | 321.9 (106.6) | 331.1 (121.7)
  PO/NG Cyclosporine dose, 12 months PT (n=170, 170) | 294.7 (93.8) | 305.7 (116.6)
  Cumulative corticosteroids,6 months PT(n=203, 206) | 848.1 (402) | 955.4 (442.8)
  Cumulative corticosteroids,12 months PT(n=195,200) | 1199.6 (771.8) | 1288.9 (796.1)

9. Secondary Outcome: Median Change From Baseline for Lipid Profile (Total Cholesterol, Low Density Lipoproteins, High Density Lipoproteins, and Triglycerides)
Description: Lipid profile included total cholesterol, low density lipoproteins (LDL), high density lipoproteins (HDL), and triglycerides (all total cholesterol, LDL, HDL, and triglycerides with unit milligram per decilitre [mg/dL]), were reported. The median change from baseline (Day -2) in lipid profile values at 3 months and 6 months was reported.
Time Frame: From Baseline (Day -2) to 3 months and 6 months
Population: The randomized population included all participants who were randomized into the study, whether they received the study drug or not. The number of participants analyzed for the specified parameters are denoted by 'n'.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 126 | 130
mg/dL
  Total cholesterol, change at 3 months (n=119,119) | 0.65 [-3.23 to 5.69] | 0.91 [-2.20 to 4.53]
  Total cholesterol, change at 6 months (n=126,130) | 0.28 [-3.75 to 6.59] | 0.61 [-2.72 to 6.39]
  LDL, Change at 3 months (n=92,89) | 0.25 [-3.35 to 4.84] | 0.34 [-2.47 to 3.48]
  LDL, Change at 6 months (n=91,99) | 0.03 [-2.86 to 3.98] | 0.21 [-2.70 to 3.48]
  HDL, change at 3 months (n=97, 101) | 0.34 [-1.27 to 1.72] | 0.31 [-1.48 to 1.64]
  HDL, change at 6 months (n=102,112) | 0.23 [-1.53 to 1.69] | 0.20 [-1.30 to 1.17]
  Triglycerides,change at 3 months (n=104,108) | 0.26 [-9.42 to 3.71] | 0.46 [-12.5 to 7.84]
  Triglycerides,change at 6 months (n=109,117) | 0.20 [-6.48 to 8.48] | 0.44 [-11.3 to 7.21]
  LDL/HDL ratio,change at 3 months (n=91,89) | -0.44 [-4.33 to 9.41] | -0.12 [-6.73 to 3.53]
  LDL/HDL ratio,change at 6 months (n=91, 99) | -0.50 [-4.45 to 3.83] | -0.14 [-6.01 to 2.90]

10. Secondary Outcome: Median Change From Baseline for LDL/HDL Ratio
Time Frame: From Baseline (Day -2) to 3 months, and 6 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: ratio
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 91 | 99
ratio
  LDL/HDL ratio,change at 3 months (n=91,89) | -0.44 [-4.33 to 9.41] | -0.12 [-6.73 to 3.53]
  LDL/HDL ratio,change at 6 months (n=91, 99) | -0.50 [-4.45 to 3.83] | -0.14 [-6.01 to 2.90]

11. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities: Hematology Parameters
Description: A marked reference range was predefined by Roche. The marked reference range is broader than the standard reference range. Values falling outside the marked reference range (low or high) that also represent a defined change from Baseline were considered marked laboratory abnormalities (i.e. potentially clinically relevant). Hematology included hemoglobin, hematocrit, white blood cell count (WBC) with differential (including granulocytes or neutrophils, basophils, eosinophils, monocytes, lymphocytes), platelets, and erythrocyte count
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one dose of study drug (daclizumab or placebo) or commercially available daclizumab and have at least one post-baseline safety assessment (eg. any laboratory data, adverse event, etc). The number of participants analyzed for the specified parameters are denoted by 'n'.
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 210 | 204
participants
  Hematocrit-high (n=210, 203) | 0 | 0
  Hematocrit-low (n=210, 203) | 116 | 117
  Hemoglobin-high (n=210, 204) | 0 | 0
  Hemoglobin-low (n=210, 204) | 107 | 112
  Platelets-high (n=210, 203) | 2 | 1
  Platelets-low (n=210, 203) | 30 | 22
  RBC-high (n=209, 203) | 1 | 2
  RBC-low (n=209, 203) | 116 | 106
  Basophils-high (n=199, 195) | 4 | 4
  Eosinophils-high (n=199, 195) | 0 | 0
  Lymphocytes-high (n=199, 198) | 2 | 2
  Lymphocytes-low (n=199, 198) | 157 | 157
  Monocytes-high (n=199, 198) | 5 | 6
  Monocytes-low (n=199, 198) | 14 | 20
  Neutrophils-low (n= 199, 198) | 33 | 33
  WBC-high (n=207, 201) | 61 | 57
  WBC-low (n=207, 201) | 43 | 29

12. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities: Biochemistry Parameters
Description: A marked reference range was predefined by Roche. The marked reference range is broader than the standard reference range. Values falling outside the marked reference range (low or high) that also represent a defined change from Baseline were considered marked laboratory abnormalities (i.e. potentially clinically relevant). Biochemistry included blood urea nitrogen, creatinine, serum glutamic oxalacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), gamma-glutamyl transferase (GGT), phosphorous, total bilirubin, direct bilirubin, total protein, albumin, glucose, alkaline phosphatase, low density lipoprotein (LDH), uric acid, carbon dioxide, magnesium, sodium, potassium, chloride, calcium, LDL, HDL, total cholesterol, and triglycerides.
Time Frame: Up to 12 months
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 210 | 204
participants
  SGPT-high (n=200, 200) | 48 | 45
  ALP-high (n=201, 200) | 15 | 7
  SGOT-high (n=201, 200) | 22 | 25
  GGT-high (n=180, 175) | 90 | 74
  LDH-high (n=194, 191) | 53 | 54
  Total bilirubin-high (n=201, 200) | 28 | 20
  BUN-high (n= 210, 200) | 93 | 95
  Creatinine-high (n=211, 203) | 66 | 64
  Albumin-low (n=198,197) | 47 | 50
  Total protein-high (n=195,196) | 5 | 0
  Total protein-low(n=195,196) | 85 | 79
  Cholesterol-high (n=174, 174) | 3 | 4
  Triglycerides-high (n=164, 164) | 35 | 30
  Carbondioxide-high (n=206, 197) | 27 | 21
  Carbondioxide-low (n=206, 197) | 12 | 5
  Chloride-high (n=211, 203) | 1 | 3
  Chloride-low (n=211, 203) | 42 | 36
  Potassium-high (n=211, 204) | 7 | 7
  Potassium-low (n=211, 204) | 4 | 2
  Sodium-high (n=211, 203) | 2 | 1
  Sodium-low (n=211, 203) | 8 | 11
  Calcium-low (n=207, 201) | 39 | 44
  Glucose fasting-high (n=210, 203) | 28 | 27
  Glucose fasting-low (n=210, 203) | 3 | 3
  Phosphate-high (n=199, 194) | 54 | 48
  Phosphate-low (n=199,194) | 32 | 26
  Uric acid high (n=191, 188) | 23 | 20

13. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Event, and Adverse Events Leading to Premature Withdrawal
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions which worsened during this study were reported as AEs. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to 12 months
Population: Safety population included all participants who received at least one dose of study drug (daclizumab or placebo) or commercially available daclizumab and have at least one post-baseline safety assessment (eg. any laboratory data, adverse event, etc).
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 207
participants
  Any AEs | 214 | 207
  Any SAE's | 108 | 102
  Any AEs leading to premature discontinuation | 14 | 11

14. Secondary Outcome: Number of Participants With Malignancies and Opportunistic Infections
Description: The opportunistic infections included infections with Cytomegalovirus, Aspergillus, Candida, Pneumocystis, Cryptococcus, Listeria, Herpes simplex, Herpes zoster. For malignancy, participants with any type of malignancy whose date of onset or diagnosis was after randomization was reported.
Time Frame: Up to 12 months
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Daclizumab | Placebo
Number analyzed (Participants) | 216 | 207
participants
  Participants with malignancies | 11 | 11
  Participants with opportunistic infections | 71 | 80

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Safety population included all participants who received at least one dose of study drug (daclizumab or placebo) or commercially available daclizumab and have at least one post-baseline safety assessment (eg. any laboratory data, adverse event, etc). The number of participants analyzed for the specified parameters are denoted by 'n'.
Arm/Group | Daclizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 108/216 | 102/207
Other Adverse Events (participants affected / at risk) | 210/216 | 204/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daclizumab (N=216) | Placebo (N=207)
Coagulation disorder nos (Blood and lymphatic system disorders) | 1 | 0
Leukopenia nos (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia nos (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 2 | 5
Atrial tachycardia (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block nos (Cardiac disorders) | 1 | 0
Bradycardia nos (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 6 | 7
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac failure nos (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 3 | 3
Cardiogenic shock (Cardiac disorders) | 2 | 0
Coronary artery disease nos (Cardiac disorders) | 0 | 1
Endocarditis nos (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 6 | 4
Post myocardial infarction syndrome (Cardiac disorders) | 0 | 1
Pulmonary oedema nos (Cardiac disorders) | 0 | 2
Right ventricular failure (Cardiac disorders) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia nos (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular arrhythmia nos (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Antibiotic associated colitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Caecum perforation (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Food poisoning nos (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis nos (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage nos (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage nos (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Mesenteric occlusion (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation nos (Gastrointestinal disorders) | 0 | 1
Toxic dilatation of colon (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Debility (General disorders) | 1 | 1
Heparin-induced thrombocytopenia nos (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 4
Pyrexia (General disorders) | 4 | 3
Sudden cardiac death (General disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Humoral immune defect (Immune system disorders) | 1 | 0
Abscess nos (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Clostridial infection nos (Infections and infestations) | 0 | 1
Empyema nos (Infections and infestations) | 1 | 0
Gastroenteritis nos (Infections and infestations) | 1 | 1
Gastroenteritis viral nos (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Injection site infection (Infections and infestations) | 2 | 0
Interstitial pneumonia (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pleural infection nos (Infections and infestations) | 1 | 0
Pneumonia gram-negative bacterial nos (Infections and infestations) | 1 | 0
Pneumonia nos (Infections and infestations) | 6 | 5
Purulent pericarditis (Infections and infestations) | 1 | 0
Sepsis nos (Infections and infestations) | 7 | 4
Septic shock (Infections and infestations) | 2 | 0
Septicaemia staphylococcal (Infections and infestations) | 0 | 1
Septicaemia streptococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection nos (Infections and infestations) | 2 | 0
Urinary tract infection nos (Infections and infestations) | 0 | 2
Viral infection nos (Infections and infestations) | 2 | 1
Wound infection nec (Infections and infestations) | 6 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 2 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Post procedural drainage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Postoperative haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Therapeutic agent poisoning (Injury, poisoning and procedural complications) | 0 | 1
Traumatic chest injury nos (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture nos (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 2
Liver function tests nos abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus nos (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 4 | 3
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia nos (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenoma benign nos (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Precancerous skin lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 2 | 1
Compartment syndrome (Nervous system disorders) | 0 | 1
Convulsions nos (Nervous system disorders) | 4 | 1
Encephalopathy nos (Nervous system disorders) | 2 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 2
Headache nos (Nervous system disorders) | 1 | 0
Intracranial haemorrhage nos (Nervous system disorders) | 2 | 0
Migraine nos (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression nos (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Calculus renal nos (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Loin pain (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 8
Renal failure nos (Renal and urinary disorders) | 2 | 3
Renal impairment nos (Renal and urinary disorders) | 2 | 3
Renal tubular necrosis (Renal and urinary disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumothorax nos (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Arterial haemorrhage nos (Vascular disorders) | 1 | 0
Cerebellar infarction (Vascular disorders) | 0 | 1
Cerebral haemorrhage (Vascular disorders) | 1 | 0
Cerebral infarction (Vascular disorders) | 1 | 2
Cerebrovascular accident nos (Vascular disorders) | 0 | 1
Deep venous thrombosis nos (Vascular disorders) | 1 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haemorrhage nos (Vascular disorders) | 0 | 1
Hypertension nos (Vascular disorders) | 0 | 1
Hypotension nos (Vascular disorders) | 0 | 2
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 0 | 2
Lymphorrhoea (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral vascular disorder nos (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
Pulmonary hypertension nos (Vascular disorders) | 2 | 2
Shock (Vascular disorders) | 0 | 1
Venous thrombosis deep limb (Vascular disorders) | 1 | 2
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Excessive bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daclizumab (N=216) | Placebo (N=207)
Anaemia nos (Blood and lymphatic system disorders) | 64 | 52
Leukocytosis (Blood and lymphatic system disorders) | 15 | 16
Leukopenia nos (Blood and lymphatic system disorders) | 32 | 22
Neutropenia (Blood and lymphatic system disorders) | 17 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 26
Arrhythmia nos (Cardiac disorders) | 10 | 12
Atrial fibrillation (Cardiac disorders) | 22 | 20
Bradycardia nos (Cardiac disorders) | 16 | 17
Nodal arrhythmia (Cardiac disorders) | 19 | 17
Pericardial effusion (Cardiac disorders) | 34 | 35
Pericardial rub (Cardiac disorders) | 10 | 12
Right ventricular failure (Cardiac disorders) | 13 | 13
Supraventricular tachycardia (Cardiac disorders) | 17 | 11
Tachycardia nos (Cardiac disorders) | 10 | 11
Tricuspid valve incompetence (Cardiac disorders) | 18 | 15
Ventricular hypokinesia (Cardiac disorders) | 11 | 14
Ventricular tachycardia (Cardiac disorders) | 11 | 10
Abdominal distension (Gastrointestinal disorders) | 13 | 9
Abdominal pain nos (Gastrointestinal disorders) | 17 | 21
Abdominal pain upper (Gastrointestinal disorders) | 4 | 12
Constipation (Gastrointestinal disorders) | 81 | 80
Diarrhoea nos (Gastrointestinal disorders) | 51 | 42
Dyspepsia (Gastrointestinal disorders) | 16 | 17
Gastrointestinal upset (Gastrointestinal disorders) | 12 | 5
Hiccups (Gastrointestinal disorders) | 11 | 12
Nausea (Gastrointestinal disorders) | 88 | 101
Pharyngolaryngeal pain (Gastrointestinal disorders) | 14 | 10
Vomiting nos (Gastrointestinal disorders) | 42 | 38
Chest pain (General disorders) | 17 | 22
Fatigue (General disorders) | 36 | 43
Oedema lower limb (General disorders) | 58 | 60
Oedema nos (General disorders) | 36 | 35
Oedema peripheral (General disorders) | 18 | 19
Pain nos (General disorders) | 18 | 13
Pyrexia (General disorders) | 26 | 22
Rigors (General disorders) | 15 | 10
Weakness (General disorders) | 30 | 24
Bronchitis nos (Infections and infestations) | 7 | 12
Nasopharyngitis (Infections and infestations) | 16 | 10
Pneumonia nos (Infections and infestations) | 12 | 6
Upper respiratory tract infection nos (Infections and infestations) | 21 | 9
Urinary tract infection nos (Infections and infestations) | 18 | 12
Post procedural pain (Injury, poisoning and procedural complications) | 106 | 105
Wound secretion (Injury, poisoning and procedural complications) | 15 | 12
Liver function tests nos abnormal (Investigations) | 12 | 12
Weight increased (Investigations) | 14 | 7
Diabetes mellitus nos (Metabolism and nutrition disorders) | 7 | 12
Gout (Metabolism and nutrition disorders) | 13 | 18
Hyperglycaemia nos (Metabolism and nutrition disorders) | 58 | 72
Hyperkalaemia (Metabolism and nutrition disorders) | 29 | 22
Hyperlipidaemia nos (Metabolism and nutrition disorders) | 11 | 9
Hypervolaemia (Metabolism and nutrition disorders) | 14 | 8
Hypoglycaemia nos (Metabolism and nutrition disorders) | 15 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 12
Metabolic acidosis nos (Metabolism and nutrition disorders) | 11 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 33
Muscle cramps (Musculoskeletal and connective tissue disorders) | 21 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 11
Pain in limb (Musculoskeletal and connective tissue disorders) | 18 | 20
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 9 | 16
Dizziness (excl vertigo) (Nervous system disorders) | 42 | 32
Headache nos (Nervous system disorders) | 64 | 58
Hypoaesthesia (Nervous system disorders) | 14 | 13
Paraesthesia (Nervous system disorders) | 14 | 20
Tremor (Nervous system disorders) | 62 | 67
Agitation (Psychiatric disorders) | 23 | 12
Anxiety nec (Psychiatric disorders) | 28 | 42
Confusion (Psychiatric disorders) | 15 | 11
Depression nos (Psychiatric disorders) | 22 | 18
Insomnia (Psychiatric disorders) | 82 | 81
Dysuria (Renal and urinary disorders) | 9 | 16
Oliguria (Renal and urinary disorders) | 26 | 28
Renal impairment nos (Renal and urinary disorders) | 50 | 43
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 22 | 22
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 24
Dyspnoea nos (Respiratory, thoracic and mediastinal disorders) | 27 | 24
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 55 | 41
Pneumothorax nos (Respiratory, thoracic and mediastinal disorders) | 13 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 13
Acne nos (Skin and subcutaneous tissue disorders) | 13 | 10
Pressure sore (Skin and subcutaneous tissue disorders) | 12 | 12
Rash nos (Skin and subcutaneous tissue disorders) | 17 | 20
Hypertension nos (Vascular disorders) | 119 | 131
Hypotension nos (Vascular disorders) | 41 | 36
Pulmonary hypertension nos (Vascular disorders) | 22 | 12
Fluid overload (Metabolism and nutrition disorders) | 43 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.